CLINICAL TRIAL: NCT05210751
Title: Investigation of the Relationship Between Dual Task With Physical and Psychosocial Factors in Female Patients With Fibromyalgia
Brief Title: Dual Task in Female Patients With Fibromyalgia
Status: Completed | Type: Observational
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ilknur Naz, Assoc. Prof, Izmir Katip Celebi University
Other Study IDs: FM111
Record Dates: First submitted 2022-01-13; First posted 2022-01-27 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Fibromyalgia; Dual Task; Physical Function; Psychosocial Problem
Keywords: Fibromyalgia; dual task; physical function; Psychosocial Problem
MeSH Terms: conditions — Fibromyalgia | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women patients with fibromyalgia: women with fibromyalgia beween age 30-75
  Interventions: Other: Physical and psychosocial assessments
- Control group: Healthy female volunteers aged 30-75 years
  Interventions: Other: Physical and psychosocial assessments

INTERVENTIONS:
Other: Physical and psychosocial assessments — Dual Task Test, 6 min Walking Test, the Baecke Habitual Physical Activity Questionnaire, Multidimensional Fatigue Inventory-20, Tracking Test, General Self-Efficacy Scale the Toronto Alexithymia Scale, the Revised FM Impact Questionnaire, the Social Support Scale.

SUMMARY:
The aim of our study is to examine the relationship between dual task and physical and psychosocial factors in female patients with fibromyalgia.

We will perform Dual Task Test, 6 min Walking Test, the Baecke Habitual Physical Activity Questionnaire, Multidimensional Fatigue Inventory-20, Tracking Test, General Self-Efficacy Scale the Toronto Alexithymia Scale, the Revised FM Impact Questionnaire, the Social Support Scale.

DETAILED DESCRIPTION:
Dual-tasking is a procedure that requires an individual to perform two tasks simultaneously to compare performance with single-task conditions, and the characteristics associated with dual-task performance in patients with fibromyalgia are unclear. Therefore, in our study, we focused on examining the relationship between dual task and physical and psychosocial factors.

Patients with a diagnosis of fibromyalgia will be included in our study.

Dual-task assessment of women with FM is with the "Dual Task Test", aerobic capacity with the "6 min Walking Test", physical activity level with the "Baecke Habitual Physical Activity Questionnaire", fatigue levels with the "Multidimensional Fatigue Inventory-20", cognitive levels With the "Tracking Test", self-efficacy levels with the "General Self-Efficacy Scale", alexithymia levels with the "Toronto Alexithymia Scale", quality of life with the "Revised FM Impact Questionnaire", motivation levels with the "Social Support Scale" will be evaluated .

ELIGIBILITY:
Inclusion Criteria:

* Women aged 30-75 years
* Patients diagnosed with fibromyalgia by a rheumatologist according to criteria set by the American College of Rheumatology
* Patients who can communicate effectively with study staff.
* Patients who have read, understood and signed the informed consent form

Exclusion Criteria:

* Those who are pregnant
* Participants who could not sit and stand in a chair even once, or climb stairs unaided
* Other rheumatic diseases and other severe somatic or psychiatric disorders such as cancer, severe coronary disease, or other serious somatic or psychiatric disorders such as schizophrenia

Ages: 30 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: - Women Women Patients aged 30-75 years diagnosed with fibromyalgia by a rheumatologist according to criteria set by the American College of Rheumatology and healthy control group
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Dual Task Assessment | 5 minutes
  Timed Up and Go Test: Participants are required to get up from the chair without assistance from their arms, walk 3 meters as fast as possible without running, turn their backs, walk back to the chair, and sit without assistance from their arms. The dual-task condition is performed by counting aloud backwards by twos, starting with a random number greater than 100 while performing the tests. Test result is saved in seconds

SECONDARY OUTCOMES:
Functional capacity | 15 minutes
  Six minute walk tests: Patients are asked to walk as fast as possible at their own walking pace for 6 minutes on a 30-meter straight corridor. At the end of the test, the walking distance is recorded.
Physical Activity Assessment | 15 minutes
  Baecke Habitual Physical Activity Questionnaire (BPAQ): The BPAQ is a self-report questionnaire to assess routine physical activity. The Baecke questionnaire is a tool that evaluates individual's habitual physical activities over the previous 12 months. This questionnaire consists of 16 questions within three main domains of individual physical activities (occupational, sport, and recreational), in the previous 12 months. Measurement of individual physical activities is achieved by calculating the sum of the scores obtained from occupational, sport, and recreational categories
Fatigue Assessment | 10 minutes
  Multidimensional Fatigue Inventory-20 (MPI): Evaluates 5 dimensions of fatigue: general fatigue, physical fatigue, mental fatigue, motivation and activity. MPI consists of 20 questions in total, with 4 questions in each subscale. Questions score between 1 and 5. The score of each subscale ranges from 4 (best) to 20 (worst).
Self-Efficacy Assessment | 10 minutes
  General Self-Efficacy Scale: The scale is a 10-item Likert-type four-point scale (1= not suitable for me at all, 2= somewhat suitable for me, 3= mostly suitable for me, 4= completely suitable for me). All items in the scale included positive statements, and those who participated in the scale were asked to answer each item using ratings ranging from "totally suitable for me" to "not at all suitable for me".
Alexithymia Assessment | 15 minutes
  Toronto Alexithymia Scale: Toronto Alexithymia Scale (TAS-20), a 20-item Likert-type self-rating scale, scored between 1-5 as "1=never" and "5=always", "Difficulty Recognizing Emotions", "Speaking Emotions" It consists of three subscales: Difficulty in Pouring and Expressive Thinking. The Difficulty Recognizing Emotions subscale consisted of seven items (items 1, 3, 6, 7, 9, 13, 14); The Difficulty in Expressing Emotions subscale includes five items (items 2, 4, 11, 12, 17) and the Expressive Thinking subscale includes eight items (items 5, 8, 10, 15, 16, 18, 19, 20). Items 4, 5, 10, 18 and 19 are scored in reverse order. High scores from the scale indicate a high level of alexithymia.
Fibromyalgia Impact Assessment | 20 minutes
  Revised Fibromyalgia Impact Questionnaire: The revised Fibromyalgia Impact Questionnaire is a questionnaire that evaluates the limitations and functional disability of patients with fibromyalgia with a total of 21 questions in three sections: function, general and symptoms. All questions are evaluated on a numerical scale between 0-10. A score of 70 and above indicates severe disability in this patient group. The higher the score obtained from the questionnaire, the higher the disability due to fibromyalgia.
Assessment of Social Support | 20 minutes
  Medical Outcome Study Social Support Scale (MOS-SSS): The first item assesses the number of close relatives and friends (structural social support). The remaining 19 items of the test are answered on a 5-point Likert-type scale ranging from 1 (never) to 5 (always). The test consists of four sub-dimensions: emotional-informational support (8 items), positive interaction (3 items), love support (4 items), and concrete support (3 items).
Cognitive Assessment | 20 minutes
  Trail Making Test: This test evaluates attention speed, mental flexibility, visual scanning and motor-speed. In part A, points 1-25 are combined with a single continuous line, in part B, a letter is combined with a number alternately. Part B has also been reported to be an indicator of executive functions. In the evaluation of the test, time and error numbers were used in the literature, but it was also reported that only the time could be used with the effect of the error on the time score by returning the last item without error to the last point reached without error. In our study, this method will be followed and only time scores will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- İlknur Naz Gürşan, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No